CLINICAL TRIAL: NCT06040697
Title: Formative Usability Assessment of Wireless Thermal Anisotropy Devices Measuring Flow in Cerebrospinal Fluid Shunts
Brief Title: Formative Usability Assessment of Wireless Thermal Anisotropy Devices
Status: Recruiting | Type: Observational
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-02
Record Dates: First submitted 2023-08-31; First posted 2023-09-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Usability Assessment Cohort: No interventions administered. Device usability assessment only.
  Interventions: Device: Thermal Anisotropy

INTERVENTIONS:
Device: Thermal Anisotropy — Usability assessment observation.
  Other Names: FlowSense

SUMMARY:
Measurements of shunt flow will be performed non-invasively. This study will generate usability data via observed tasks and comprehension questions to enable future device design improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Existing ventricular CSF shunt with a region of intact skin overlying the shunt catheter appropriate in size for application of the study device
2. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
3. Subject or caregiver can clearly communicate and document information in English
4. Verbal assent by minors 12 years of age and older who can understand the study and communicate their decision
5. Subject is at least 5 years old but not more than 80 years old

Exclusion Criteria:

1. Presence of an interfering open wound in the device application region
2. Subject-reported history of adverse skin reactions to adhesives

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with an existing Cerebrospinal Fluid (CSF) shunt
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Exploratory device usability feedback | 2 hours
  Identification of usability risks [unscored]

CONTACTS AND LOCATIONS:
Locations (1):
- Rhaeos, Inc., Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No